CLINICAL TRIAL: NCT00298428
Title: Biological Efficacy of Clopidogrel 600 mg Loading Dose Followed by 75 mg Maintenance Dose After Implantation of Drug-eluting Stents in Patients With Diabetes Mellitus or Metabolic Syndrome (SPACE)
Brief Title: Biological Efficacy of Clopidogrel After Implantation of Drug-eluting Stents (SPACE)
Acronym: SPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P051004
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Diabetes Mellitus; Metabolic Syndrome X
Keywords: stent; percutaneous coronary intervention; platelet aggregation; clopidogrel; shear; metabolic syndrome
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Diabetes Mellitus; Metabolic Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPACE group (Other)
  Interventions: Procedure: blood samples

INTERVENTIONS:
Procedure: blood samples — blood samples before percutaneous coronary intervention (PCI) and at 4 months
  Other Names: blood samples before percutaneous coronary intervention

SUMMARY:
The risk of thrombotic complications after implantation of drug-eluting stents (DES) may be increased in patients with diabetes mellitus (DM) or metabolic syndrome (MS). It is recommended that all patients take an association of aspirin and clopidogrel for several months after DES implantation to reduce this risk. However, the biological efficacy of current antiplatelet therapies has not been studied prospectively and specifically in DM or MS patients.

Our aim is to study the biological efficacy of an association of aspirin and clopidogrel (600 mg loading dose followed by 75 mg maintenance dose) using an assay measuring ex vivo shear-induced platelet aggregation (SIPA), along with other assays measuring platelet activation and aggregation, in patients with DM, MS, or no DM/MS.

Patients with stable coronary artery disease and successful DES implantation in native coronary arteries will be eligible. They will be stratified at entry according to their metabolic status (DM, MS, or no DM/MS). Measurements will be performed 6-24 hours after clopidogrel loading dose (acute effects) and 4 months later under clopidogrel maintenance dose (chronic effects).

Study end-points:

A. Primary biological end-point: To compare SIPA levels in DM vs. MS vs. no DM/MS patients.

B. Secondary biological end-points:

* To compare the results of other tests of platelet aggregation/activation in DM vs. MS vs. no DM/MS patients.
* To compare the acute (6-24 hours after clopidogrel loading dose) and chronic (4 months later) results of the above mentioned tests. These comparisons will be performed in the overall population and in each group (DM, MS, no DM/MS).

C. Secondary clinical end-points: To study the relationship between SIPA levels (and the other tests of platelet aggregation/activation) and the occurrence of:

* Periprocedural myocardial infarctions
* Major adverse cardiac events (cardiovascular death, myocardial infarction or ischaemia-driven target vessel revascularization) at 4 and 12 months after stent implantation.

We, the researchers at Assistance PUBLIQUE - HOPITAUX de Paris, anticipate our study may help improve our knowledge of the efficacy of current antiplatelet therapies in DM and MS patients treated with DES.

DETAILED DESCRIPTION:
The risk of thrombotic complications after implantation of drug-eluting stents (DES) in coronary arteries may be increased in patients with diabetes mellitus (DM) or metabolic syndrome (MS). It is recommended that all patients take an association of aspirin and clopidogrel for several months after DES implantation to reduce this risk. However, the biological efficacy of current antiplatelet therapies has not been studied prospectively and specifically in DM or MS patients.

In the present study, we will study the biological efficacy of an association of aspirin and clopidogrel (600 mg loading dose followed by 75 mg maintenance dose) using an assay measuring ex vivo shear-induced platelet aggregation (SIPA), along with other assays measuring platelet activation and aggregation, in order to better describe the heterogeneity of response to antiplatelet agents in patients with DM, MS or no DM/MS.

All patients with stable coronary artery disease and successful DES implantation in native coronary arteries (including high risk features, eg, left main stenosis, bifurcations or in-stent restenosis) will be eligible. They will be stratified at entry according to their metabolic status (DM, MS, or no DM/MS). Measurements will be performed both 6-24 hours after clopidogrel loading dose (acute effects) and 4 months later under clopidogrel maintenance dose (chronic effects).

Study end-points:

A. Primary biological end-point: To compare SIPA levels in DM vs. MS vs. no DM/MS patients.

B. Secondary biological end-points:

* To compare the results of other tests of platelet aggregation/activation (light transmittance aggregometry in response to ADP and arachidonic acid; flow cytometry measurements of VASP phosphorylation, platelet expression of P-selectin and GPIIbIIIa, and circulating levels of platelet microparticles and leukocyte-platelet aggregates; PFA-100 occlusion time; circulating levels of thromboxane B2) and circulating levels of other markers of atherosclerosis (CRPhs, von Willebrand factor, PAI-1, fibrinogen, and soluble CD40L) in DM vs. MS vs. no DM/MS patients.
* To compare the acute (6-24 hours after clopidogrel loading dose) and chronic (4 months later) results of all the above mentioned tests. These comparisons will be performed in the overall population and in each group (DM, MS, no DM/MS).

C. Secondary clinical end-points: To study the relationship between SIPA levels (and the other tests of platelet aggregation/activation) and the occurrence of:

* Periprocedural myocardial infarctions
* Major adverse cardiac events (cardiovascular death, myocardial infarction or ischaemia-driven target vessel revascularization) at 4 and 12 months after stent implantation.

We anticipate our study may help improve our knowledge of the efficacy of current antiplatelet therapies in DM and MS patients treated with DES.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented myocardial ischaemia (stable angina with positive stress ECG or stress myocardial scintigraphy, silent ischemia with positive stress ECG or stress myocardial scintigraphy, non-ST elevation acute coronary syndrome)
* Treatment with at least 100 mg/day of aspirin for ≥ 6 hours before percutaneous coronary intervention
* 600 mg clopidogrel loading-dose given ≥ 6 hours and < 24 hours before coronary angiography
* Presence of one or several stenosis in native coronary arteries requiring percutaneous coronary intervention and implantation of one or several drug-eluting stents

Exclusion Criteria:

* ST-elevation acute coronary syndrome
* Pregnancy or breast feeding
* Severe disease with life expectancy lower than 1 year
* High bleeding risk (blood coagulation disorders, uncontrolled severe hypertension, active bleeding, history of severe bleeding)
* Intolerance or contraindication to aspirin or clopidogrel
* Current treatment (or stopped < 10 days) with vitamin K antagonist
* Current treatment (or stopped < 10 days) with clopidogrel (except for the clopidogrel loading-dose given prior to percutaneous coronary intervention), ticlopidine, dipyridamole, non-steroidal antiinflammatory agent, GPIIB-IIIA blocker
* One-year follow-up impossible
* Refusal to sign the information and consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Primary biological end-point: To compare SIPA levels in DM vs. MS vs. no DM/MS patients | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent J Feldman, MD, PhD, Principal Investigator — Département de Cardiologie, Hôpital Bichat, Assistance Publique-Hôpitaux de Paris; Nadine Ajzenberg, MD, PhD, Principal Investigator — Service d'Hématologie et d'Immunologie Biologiques, Hôpital Bichat, Assistance Publique-Hôpitaux de Paris
Locations (2):
- France (2):
  - Département de Cardiologie, Hôpital Bichat, Assistance Publique-Hôpitaux de Paris, Paris
  - Service d'Hématologie et d'Immunologie Biologiques, Hôpital Bichat, Assistance Publique-Hôpitaux de Paris, Paris

REFERENCES:
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Serebruany VL, Steinhubl SR, Berger PB, Malinin AI, Bhatt DL, Topol EJ. Variability in platelet responsiveness to clopidogrel among 544 individuals. J Am Coll Cardiol. 2005 Jan 18;45(2):246-51. doi: 10.1016/j.jacc.2004.09.067. PMID 15653023
- [Background] Gurbel PA, Bliden KP, Hiatt BL, O'Connor CM. Clopidogrel for coronary stenting: response variability, drug resistance, and the effect of pretreatment platelet reactivity. Circulation. 2003 Jun 17;107(23):2908-13. doi: 10.1161/01.CIR.0000072771.11429.83. Epub 2003 Jun 9. PMID 12796140
- [Background] Kastrati A, Mehilli J, Schuhlen H, Dirschinger J, Dotzer F, ten Berg JM, Neumann FJ, Bollwein H, Volmer C, Gawaz M, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic Regimen-Rapid Early Action for Coronary Treatment Study Investigators. A clinical trial of abciximab in elective percutaneous coronary intervention after pretreatment with clopidogrel. N Engl J Med. 2004 Jan 15;350(3):232-8. doi: 10.1056/NEJMoa031859. PMID 14724302
- [Background] Patti G, Colonna G, Pasceri V, Pepe LL, Montinaro A, Di Sciascio G. Randomized trial of high loading dose of clopidogrel for reduction of periprocedural myocardial infarction in patients undergoing coronary intervention: results from the ARMYDA-2 (Antiplatelet therapy for Reduction of MYocardial Damage during Angioplasty) study. Circulation. 2005 Apr 26;111(16):2099-106. doi: 10.1161/01.CIR.0000161383.06692.D4. Epub 2005 Mar 6. PMID 15750189
- [Background] Matetzky S, Shenkman B, Guetta V, Shechter M, Beinart R, Goldenberg I, Novikov I, Pres H, Savion N, Varon D, Hod H. Clopidogrel resistance is associated with increased risk of recurrent atherothrombotic events in patients with acute myocardial infarction. Circulation. 2004 Jun 29;109(25):3171-5. doi: 10.1161/01.CIR.0000130846.46168.03. Epub 2004 Jun 7. PMID 15184279
- [Background] Ajzenberg N, Aubry P, Huisse MG, Cachier A, El Amara W, Feldman LJ, Himbert D, Baruch D, Guillin MC, Steg PG. Enhanced shear-induced platelet aggregation in patients who experience subacute stent thrombosis: a case-control study. J Am Coll Cardiol. 2005 Jun 7;45(11):1753-6. doi: 10.1016/j.jacc.2004.10.079. PMID 15936600